CLINICAL TRIAL: NCT00127920
Title: A Phase II, Open-Label, Non-Randomized, Multi-Center Pilot Study of Intravenous Taxol, Carboplatin, Bevacizumab Given Every 21 Days in Patients With Newly Diagnosed Stage III/IV Epithelial Ovarian, Fallopian Tube or Peritoneal Cancer
Brief Title: Pilot Study of Taxol, Carboplatin, and Bevacizumab in Advanced Stage Ovarian Carcinoma Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Associates (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AV53206s
Record Dates: First submitted 2005-08-05; First posted 2005-08-09 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Ovarian Neoplasms
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm (Experimental): Paclitaxel, Carboplatin and Avastin on day1 every 21 days
  Interventions: Drug: Avastin

INTERVENTIONS:
Drug: Avastin — Paclitaxel, Carboplatin and Avastin given on day 1 every 21 days
  Other Names: Bevacizumab

SUMMARY:
The most likely way to improve survival and cure rates in treating ovarian cancer, fallopian tube epithelial cancer, and peritoneal cancer is with maximal "upfront" therapy (Morrow & Curtin, 1998). This involves an optimal primary tumor debulking surgery. The most active chemotherapy agents should then be promptly administered. Taxol and Carboplatin or Cisplatin have become the standard" first line" therapy because of proven survival benefits with those regimens in treating advanced ovarian adenocarcinoma patients. New chemotherapy agents like bevacizumab have demonstrated increased overall and progression free survival benefits in metastatic colorectal cancer patients and are being studied for their potential contributory impact on the current standard of treatment. Since no triplet regimen has demonstrated compelling superiority, the combination of taxol, carboplatin, and bevacizumab is intriguing because of their potential synergy, distinct mechanisms of action, and non-overlapping toxicity.

The null hypothesis (Ho) is that the drug regimen will demonstrate an 80% patient response rate (RR).

The alternative Hypothesis (H1): The triplet drug regimen will demonstrate a significantly higher patient response rate than standard therapy.

Hypothesis (H2): The triplet drug regimen will demonstrate a significantly more favorable patient time to tumor progression rate than standard therapy.

DETAILED DESCRIPTION:
The most likely way to improve survival and cure rates in treating ovarian cancer, fallopian tube epithelial cancer, and peritoneal cancer is with maximal "upfront" therapy. This involves an optimal primary tumor debulking surgery. The most active chemotherapy agents should then be promptly administered. Taxol and Carboplatin or Cisplatin have become the standard" first line" therapy because of proven survival benefits with those regimens in treating advanced ovarian adenocarcinoma patients. New agents like bevacizumab (Avastin), which have demonstrated increased overall and progression free survival benefits in metastatic colorectal cancer patients, are being added to the optimal first line ovarian chemotherapy regimen in hopes of seeing improvement in progressive free interval and over-all survival. Since no triplet regimen has demonstrated compelling superiority, the combination of taxol, carboplatin, and bevacizumab (Avastin) is intriguing because of their potential synergy, distinct mechanisms of action, and non-overlapping toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a histologic or cytologic diagnosis of stage III/IV ovarian cancer, fallopian tube epithelial cancer, or peritoneal cancer who have not received prior chemotherapy or radiotherapy.
* Subjects must have the appropriate surgery for their gynecologic cancer. However, subjects may be treated in a neoadjuvant manner, with surgery being performed after chemotherapy cycles 1, 2, or 3.
* If neoadjuvant therapy is not administered, subjects must receive their first dose no more than six weeks postoperatively.
* Subjects must have adequate bone marrow, renal and hepatic function as defined by WBC > 3,000 cells/cu ml., platelets > 100,000/cu.ml., calculated creatinine clearance > 50 ccs/min., bilirubin < 1.5 mg/dl, and SGOT < three times normal.
* Karnofsky performance status > 50%.
* Subjects who have signed an institutional review board (IRB) approved informed consent form.

Exclusion Criteria:

* Subjects with epithelial ovarian cancer of low malignancy potential.
* Subjects with septicemia, severe infection, or acute hepatitis.
* Subjects with severe gastrointestinal bleeding.
* Subjects with a history of congestive heart failure, angina, or a history of myocardial infarction within the past six months.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2004-08; Primary Completion 2006-08 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
time to tumor progression
response rate

SECONDARY OUTCOMES:
safety
survival

CONTACTS AND LOCATIONS:
Overall Officials: John P Micha, MD, Principal Investigator — Gynecologic Oncology Associates
Locations (2):
- United States (2):
  - Gynecologic Oncology Associates, Newport Beach, California
  - Florida Hospital College of Health Sciences, Orlando, Florida